CLINICAL TRIAL: NCT01989234
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, 12-Week, Dose-Range-Finding Trial of YKP10811 Capsules Administered Once Daily to Subjects With Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YKP10811C006
Record Dates: First submitted 2013-10-30; First posted 2013-11-20 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — carbamic acid 3-(4-((4-amino-5-chloro-2-methoxybenzoylamino)methyl)piperidin-1-yl)-1-(4-fluorophenyl)propyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo Comparator (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo
- YKP10811 High Dose (Experimental): YKP10811 High Dose
  Interventions: Drug: YKP10811
- YKP10811 Mid Dose (Experimental): YKP10811 Mid Dose
  Interventions: Drug: YKP10811
- YKP10811 Low Dose (Experimental): YKP10811 Low Dose
  Interventions: Drug: YKP10811

INTERVENTIONS:
Drug: YKP10811
  Arms: YKP10811 High Dose; YKP10811 Low Dose; YKP10811 Mid Dose
Drug: Placebo
  Arms: Placebo Comparator

SUMMARY:
This will be a multi-center, randomized, double-blind, placebo-controlled study of YKP10811 capsules in patients with chronic idiopathic constipation. Following a 2-week baseline period, approximately 320 eligible patients with <3 complete spontaneous bowel movements (CSBM) and ≤ 5 SBMs per week will be randomly assigned equally to receive one of the following oral treatments; placebo or YKP10811 capsules once daily for 12 weeks followed by a 2 week follow-up period.

The objectives of this study are:

* To assess the efficacy of YKP10811 once daily at relieving constipation and associated symptoms in subjects with chronic idiopathic constipation.
* To determine the safety and tolerability of YKP10811 once daily in subjects with chronic idiopathic constipation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet modified Rome II criteria for Chronic Constipation.
* Patients who are male or female, 18 to 65 years of age inclusive.
* At Visit 3, patients must have < 3 CSBMs per week and ≤ 5 SBMs per week during the 2-week baseline period.

Exclusion Criteria:

* Patients who meet Rome II criteria for Irritable Bowel Syndrome (IBS-C).
* Patients with constipation that is drug-induced, or secondary to endocrine, metabolic or, surgery.
* Patients with a clinically significant diseases that would limit the patient's ability to complete and/or participate in the study, including gastrointestinal disorder or surgery, an endocrine abnormality (e.g., diabetes), impaired renal function (GFR of < 55mL/minute/1.73m2), uncontrolled pulmonary diseases (including asthma), uncontrolled cardiovascular disease (a history of myocardial infarction or cerebrovascular accident within 6 months prior to screening) or significant neurological diseases.
* Patients with a history of inflammatory bowel disease.
* Patients with a history of cancer (other than basal cell or squamous cell carcinoma of the skin completely excised) unless the malignancy has been in complete remission for at least 5 years prior to screening.
* Patients who started a special diet and/or an intense physical workout program within 30 days prior to the beginning of the baseline period or who are intending to substantially modify their dietary habits at any time during the study (patients on a stable, continuous regimen of fiber therapy for at least 30 days prior to the pretreatment baseline period are allowed to continue that therapy, provided that they continue at a constant dose throughout the study.
* Patients with a history of clinically significant hypersensitivity or allergy (facial swelling, hives, breathing difficulty, Stevens-Johnson syndrome etc), in response to any medication, either prescription or nonprescription including an investigational drug, dietary supplement, or herbal medicine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with improved bowel movement frequency | 12 weeks

SECONDARY OUTCOMES:
Stool frequency | 12 weeks
Daily average ratings of stool consistency | 12 weeks
Instances of rescue medicine usage | 12 weeks
Onset time to CSBM | 12 weeks
Onset time to SBM | 12 weeks
Severity of straining | 12 weeks
Abdominal discomfort | 12 weeks
Abdominal pain | 12 weeks
Bloating | 12 weeks
Constipation severity | 12 weeks

CONTACTS AND LOCATIONS:
Locations (69):
- United States (69):
  - Alliance Clinical Research, Birmingham, Alabama
  - Clinical Research Advantage, Inc. / Warner Family Practice, PC, Chandler, Arizona
  - Connect Clinical Research Center, Chandler, Arizona
  - Clinical Research Advantage, Inc. / Central Phoenix Medical Clinic, LLC, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Applied Research Center Arkansas, Inc., Little Rock, Arkansas
  - Digestive & Liver Disease Specialists, A Medical Group, Inc., Anaheim, California
  - Precision Research Institute, Chula Vista, California
  - Triwest Research Associates, LLC, El Cajon, California
  - Diagnamics Inc., Encinitas, California
  - Therapeutic Research Institute of Orange County, Laguna Hills, California
  - Clinical Trials Research, Lincoln, California
  - Alliance Clinical Research, Oceanside, California
  - Northern California Research, Sacramento, California
  - Clinical Research Advantage, Inc. / Colorado Springs Health Partners, SW, Colorado Springs, Colorado
  - Meridien Research, Bradenton, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - The Clinical Research Institute, Miami, Florida
  - Prestige Clinical Research Center Inc., Miami, Florida
  - Physicians Regional Medical Group, Naples, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - May Medical Center, Chicago, Illinois
  - Pharmakon Inc., Evergreen Park, Illinois
  - Clinical Research Advantage, Inc., Evansville, Indiana
  - KAMP Medical Research, Inc., Natchitoches, Louisiana
  - Clinical Associates Ambulatory Surgical Center, Towson, Maryland
  - The Research Institute, Springfield, Massachusetts
  - Coastal Research Associates, Inc., Weymouth, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Clinical Research Advantage, Inc., Henderson, Nevada
  - AB Clinical Trials, Las Vegas, Nevada
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Las Vegas, Nevada
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - HBSA, A Supporting Organization of Pacific Institute for Research and Evaluation, Albuquerque, New Mexico
  - NY Scientific, Brooklyn, New York
  - Medex Healthcare Research, Inc., New York, New York
  - PMG Research of Charlotte, Charlotte, North Carolina
  - PMG Research of Charlotte, Concord, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Dayton Gastroenterology, Inc., Beavercreek, Ohio
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Hilltop Physicians IN / Hightop Medical Research Center, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Columbus Clinical Research Inc., Columbus, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - The Oregon Clinic, PC - Gastroenterology West, Portland, Oregon
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Partners in Clinical Research, LLC, Cumberland, Rhode Island
  - Health Concepts, Rapid City, South Dakota
  - Alpha Clinical Research, LLC, Clarksville, Tennessee
  - Austin Center for Clinical Research, Austin, Texas
  - MW Clinical Research Center, Beaumont, Texas
  - Houston Endoscopy & Research Center, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - Radiant Research Inc., San Antonio, Texas
  - Digestive Health Specialists of Tyler, LLP, Tyler, Texas
  - Advanced Research Institute, Ogden, Utah
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia